CLINICAL TRIAL: NCT07267260
Title: Evaluating the Efficacy of Vonoprazan in Preventing Post-Endoscopic Variceal Band Ligation Ulcers: A Randomized Controlled Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Rizwan Tariq Neuro, Principal Investigator, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 640/RC/KEMU Dated: 28/08/25; 640/RC/KEMU (Other: IRB King Edward Medical University)
Record Dates: First submitted 2025-11-23; First posted 2025-12-05 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cirrhoses, Liver
Keywords: Vonoprazan; Potassium-competitive acid blocker; Endoscopic variceal band ligation; Esophageal varices; Post-procedure ulcer; Cirrhosis; Portal hypertension; Double-blind randomized controlled trial
MeSH Terms: conditions — Esophageal and Gastric Varices; Fibrosis; Hypertension, Portal | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vonoprazan 20 mg after EVBL (Experimental): Participants in this arm will receive vonoprazan 20 mg orally once daily for 14 days following endoscopic variceal band ligation (EVBL). Vonoprazan is a potassium-competitive acid blocker that provides strong and sustained suppression of gastric acid. The aim is to test whether vonoprazan can help prevent the formation of ulcers that sometimes develop after EVBL and to improve symptoms such as pain or difficulty swallowing. Participants will continue their usual medical care for liver disease. Study staff, participants, and investigators will all remain blinded to treatment allocation until data analysis is complete.
  Interventions: Drug: Vonoprazan 20 mg
- Placebo after EVBL (Placebo Comparator): Participants in this arm will receive a placebo tablet orally once daily for 14 days following endoscopic variceal band ligation (EVBL). The placebo tablet will look identical to the Vonoprazan tablet but contains no active medicine. This group serves as a comparison to determine whether Vonoprazan is more effective than placebo in preventing post-procedural ulcers and reducing symptoms such as swallowing discomfort or chest pain. Participants will receive standard medical care for liver disease and will undergo the same follow-up and assessments as the experimental group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vonoprazan 20 mg — Vonoprazan is a potassium-competitive acid blocker (P-CAB) that provides strong and sustained suppression of gastric acid secretion. In this study, participants will receive vonoprazan 20 mg by mouth once daily for 14 days after endoscopic variceal band ligation (EVBL). The tablets will be taken with water, preferably before breakfast. This dose and duration are based on prior clinical experience in acid-related disorders. The aim is to determine whether vonoprazan prevents the formation of ulcers and reduces post-procedure pain compared with placebo.
  Other Names: Potassium-competitive acid blocker; TAK-438
  Arms: Vonoprazan 20 mg after EVBL
Other: Placebo — Participants in the placebo group will receive a look-alike oral tablet with no active medicine, once daily for 14 days after EVBL. The placebo will be identical in color, size, and packaging to the Vonoprazan tablet to maintain blinding. This comparator will help determine whether Vonoprazan provides any true benefit in preventing ulcers and improving symptoms beyond standard post-procedure care.
  Other Names: Inactive tablet
  Arms: Placebo after EVBL

SUMMARY:
The goal of this clinical trial is to learn if the medicine vonoprazan can help prevent ulcers that may develop after endoscopic variceal band ligation (EVBL) in adults with liver cirrhosis. These ulcers sometimes cause pain or delayed bleeding after the procedure.

The study will also look at how well vonoprazan is tolerated and if it improves comfort after the procedure.

The main questions this study will answer are:

Does vonoprazan lower the number and severity of ulcers found on endoscopy after EVBL?

Does vonoprazan reduce swallowing pain or chest discomfort compared with placebo?

Is vonoprazan safe and well tolerated in people with liver cirrhosis?

Researchers will compare vonoprazan 20 mg once daily with a placebo (a look-alike tablet that contains no active medicine) to see if vonoprazan works better to prevent these ulcers.

Participants will:

Take vonoprazan or placebo by mouth once daily for 14 days after EVBL.

Return for a follow-up endoscopy about two weeks later to check for ulcers.

Report any symptoms such as pain, nausea, or swallowing difficulty during the study.

Adults aged 18 to 75 years with liver cirrhosis who undergo EVBL will be invited to join. Participants will be randomly assigned to one of two groups, and neither they nor the study doctors will know which treatment they receive (double-blind design).

The study will take place at Mayo Hospital, Lahore, Pakistan, over about six months.

By comparing vonoprazan to placebo, researchers hope to find a better way to protect the esophagus and stomach after EVBL, reduce post-procedure pain, and support faster recovery in people with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years (male or female)
* Diagnosis of liver cirrhosis confirmed by clinical, biochemical, or imaging findings.
* Presence of documented esophageal varices requiring endoscopic variceal band ligation (EVBL).
* Able and willing to provide written informed consent in English or Urdu.
* Willing to comply with study procedures, including taking study medication and attending follow-up endoscopy.

Exclusion Criteria:

* History of gastric or esophageal surgery
* Allergy or contraindication to vonoprazan or study drug components
* Pregnant or lactating women
* Individuals who are non-cooperative or unable to understand local languages
* Critically ill patients, including:

ICU admission Requirement for mechanical ventilation GCS < 10

* Active gastrointestinal bleeding at the time of enrollment
* Malignancy of the upper gastrointestinal tract

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-12-16 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post-Endoscopic Variceal Band Ligation (EVBL) Ulcers | At follow-up endoscopy, 14 ± 1 days after EVBL.
  The proportion of participants who develop visible post-banding ulcers detected on follow-up endoscopy. Ulcers will be assessed using the Lanza Score for gastric mucosal injury, which grades the number and severity of ulcers from 0 (no injury) to 4 (severe injury). A lower Lanza score indicates less mucosal injury. The outcome compares the rate and severity of ulcers between the vonoprazan and placebo groups.

SECONDARY OUTCOMES:
Change in Dysphagia, Odynophagia, and Retrosternal Pain Scores on Visual Analog Scale (VAS) | Baseline and 14 ± 1 days after EVBL.
  Change in symptom intensity for swallowing pain (odynophagia), difficulty swallowing (dysphagia), and chest discomfort (retrosternal pain), measured using a 100 mm Visual Analog Scale (VAS) where 0 = no pain and 100 = worst possible pain. The change from baseline to day 14 will be calculated. A ≥ 20% reduction in VAS score from baseline will be considered clinically significant.

CONTACTS AND LOCATIONS:
Locations (1):
- King Edward Medical University/Mayo Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly because this is a single-center academic study conducted at Mayo Hospital, Lahore, with a limited sample size and locally collected data. De-identified summary data and statistical analyses may be made available upon reasonable request to the principal investigator after publication of study results, in accordance with institutional and ethical committee policies.